CLINICAL TRIAL: NCT03484494
Title: Low Field Magnetic Stimulation: Imaging Biomarkers in Geriatric Bipolar Depression
Acronym: LFMSBioMGeri
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, David G. Harper, Ph.D., David Harper, PhD, Mclean Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2017P002783
Record Dates: First submitted 2018-02-22; First posted 2018-03-30 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Bipolar Disorder; Bipolar Depression; Bipolar I Disorder; Bipolar II Disorder
Keywords: Geriatric; Low Field Magnetic Stimulation; Antidepressant; fMRI; MRS
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: This is a sham controlled, randomized, double blinded crossover design study of immediate change to brain activity caused by Low Field Magnetic Stimulation.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The device is operated using subject-specific links on a laptop. The active or sham identity of the links is prepared automatically and not known to study staff or participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active first (Other): Subjects receive active Low Field Magnetic Stimulation in the first imaging visit and sham in the second.
  Interventions: Device: Low Field Magnetic Stimulation
- Sham first (Other): Subjects receive sham Low Field Magnetic Stimulation in the first imaging visit and active in the second.
  Interventions: Device: Low Field Magnetic Stimulation

INTERVENTIONS:
Device: Low Field Magnetic Stimulation — Low Field Magnetic Stimulation is an application of a series of electromagnetic pulses to the brain through a small cylinder that the subject places the top of their head inside.

SUMMARY:
The protocol involves functional Magnetic Resonance Imaging acquisitions immediately before and after Low Field Magnetic Stimulation treatment on two separate days in a sham controlled, randomized trial, in order to assess the physiologic effects of Low Field Magnetic Stimulation on brain function in a geriatric population with bipolar depression.

DETAILED DESCRIPTION:
In this study, the investigators will examine changes in brain activity from Low Field Magnetic Stimulation in subjects over the age of 50 with bipolar disorder who are currently depressed using functional Magnetic Resonance Imaging. Following screening visits, study procedures include two visits, at least two weeks apart, during which subjects will complete brief mood scales, undergo up to 15 minutes of imaging, receive 20 minutes of Low Field Magnetic Stimulation treatment, and then return to the scanner to undergo up to 15 minutes of imaging procedures. Due to the crossover design, subjects receiving active treatment during the first visit will receive sham treatment during the second visit; subjects receiving sham treatment during the first visit will receive active treatment during the second visit. A follow-up phone call will occur at least two days after each imaging/treatment visit. The main endpoint of this study is the observation of changes in resting state functional Magnetic Resonance Imaging activity in post-treatment acquisitions as compared to pre-treatment acquisitions.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will have a diagnosis of Bipolar Disorder Type I or II, current episode depressed as measure by a MADRS ≥ 20.
2. Subjects must be maintained on a stable dose of all psychotropic medications for a period of at least two weeks prior to screening.
3. Subjects must be capable of providing informed consent.
4. Subjects must permanently reside within a 2-hour drive of McLean Hospital.
5. Subjects must be currently seen by a provider (psychiatrist, therapist, PCP) whose practice is within a 2-hour drive of McLean Hospital.

Exclusion Criteria:

1. Dangerous or active suicidal ideation, as measured by the C-SSRS (see "Safety Measures" section), and physician evaluation.
2. Subjects meeting DSM-5 criteria for schizophrenia, schizoaffective disorder, or other psychotic disorders, or dementia.
3. Current mania as defined by a score of ≥ 10 on the Young Mania Rating Scale at screening.
4. Subject has an MMSE score ≤ 24.
5. Subject is pregnant or plans on becoming pregnant.
6. Subject has recent history (within 7 days of screening) of ECT or TMS treatment.
7. Subject has recent history of substance abuse (cannot meet DSM-5 criteria for substance abuse, no significant drug abuse within last 3 months, no history of dependence in last year, no drug use within last month, other than marijuana use).
8. Subject has any contraindication for MRI (i.e. Presence of a pacemaker, neurostimulator, or metal in head or neck).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-05-29 (Actual); Primary Completion 2025-05-21 (Estimated); Study Completion 2025-05-21 (Estimated)

PRIMARY OUTCOMES:
Change in resting state brain activity measured by functional Magnetic Resonance Imaging. | Resting state functional Magnetic Resonance Imaging data are acquired 4 times, twice within one hour during imaging visit 1 and twice within one hour during imaging visit 2 which occurs at least two weeks later.
  Comparison of change in brain activity occurring over the time of treatment, compared between active and sham treatment visits. This is assessed by combining pre and post treatment measures made during active and sham treatment visits using the following formula: (post active treatment - pre active treatment) - ( post sham - pre sham). The brain activity is measured using blood oxygenation level dependent image of brain activity acquired in the resting state using functional Magnetic Resonance Imaging.

CONTACTS AND LOCATIONS:
Overall Officials: David G Harper, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No